CLINICAL TRIAL: NCT02596841
Title: Lung Diffusing Capacity for Nitric Oxide as a Marker of Fibrotic Changes in Idiopathic Interstitial Pneumonias
Acronym: Dm&Vc
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy (Other)
Responsible Party: Principal Investigator, Giovanni Barisione, MD, IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy
Other Study IDs: IRCCS 2015
Record Dates: First submitted 2015-10-29; First posted 2015-11-04 (Estimated); Last update posted 2015-11-04 (Estimated); Status verified 2015-11

CONDITIONS: Usual Interstitial Pneumonia; Nonspecific Interstitial Pneumonia
Keywords: Lung diffusing capacity; Idiopathic Interstitial Pneumonias
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Idiopathic Interstitial Pneumonias

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The diagnosis of idiopathic interstitial pneumonia (IIP) is based on computed tomography (CT) imaging, whereas lung function studies are used for staging and follow up. Lung diffusing capacity for carbon monoxide (DLCO) is generally reduced but weakly correlated with the severity of CT-determined fibrotic process. A possible explanation of this finding is that DLCO is relatively insensitive to changes in alveolar membrane diffusive conductance (DMCO). Lung diffusion capacity for nitric oxide (DLNO) was strongly correlated with CT-determined amount of fibrosis/honeycombing in both usual and non-specific interstitial pneumonias. Moreover. Both DLNO and DMCO were below the lower limit of normality even in patients with small amount of fibrosis. Measurement of DLNO may provide a more reliable assessment of fibrotic changes than DLCO because it better reflects DMCO.

DETAILED DESCRIPTION:
Rationale: Lung diffusing capacity for carbon monoxide (DLCO) is decreased in both usual interstitial pneumonia-idiopathic pulmonary fibrosis (UIP-IPF) and nonspecific interstitial pneumonia (NSIP), but is weakly related to computed tomography (CT)-determined fibrotic changes.

Objectives: To determine whether measurement of lung diffusing capacity for nitric oxide (DLNO) better reflects fibrotic changes than DLCO.

Methods: DLNO and DLCO were measured simultaneously in 30 patients with UIP-IPF and 30 with NSIP. The amount of pulmonary fibrosis was estimated by volumetric analysis of visually bounded areas showing reticular opacities and honeycombing. Alveolar membrane conductance (DMCO) and pulmonary capillary volume (Vc) were calculated.

ELIGIBILITY:
Inclusion Criteria:

* Chest computed tomography (CT) scan diagnosis of either usual interstitial pneumonia-idiopathic pulmonary fibrosis (UIP-IPF) or idiopathic nonspecific interstitial pneumonia (NSIP)

Exclusion Criteria:

* Symptoms/signs or specific serum markers of an underlying autoimmune process
* Previous environmental/occupational exposure to fibrogenic dusts
* Use of fibrogenic medications

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The investigators used retrospectively collected data of 60 Caucasian patients with clinical and radiological features of Idiopathic Interstitial Pneumonias referred to Respiratory Pathophysiology Unit for a complete pulmonary function evaluation.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2013-02; Primary Completion 2015-05 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Changes of lung diffusing capacity for nitric oxide (DLNO) in a group of 60 patients with fibrosing idiopathic interstitial pneumonias (IIPs) | Within 1 month following idiopathic interstitial pneumonias diagnosis
  Because DLNO is more sensitive to alveolar membrane diffusive conductance (DMCO) than standard lung diffusing capacity for carbon monoxide, DLNO changes may better reflect the extent of fibrotic process in IIPs

REFERENCES:
- [Background] Guenard H, Varene N, Vaida P. Determination of lung capillary blood volume and membrane diffusing capacity in man by the measurements of NO and CO transfer. Respir Physiol. 1987 Oct;70(1):113-20. doi: 10.1016/s0034-5687(87)80036-1. PMID 3659606
- [Background] Borland CD, Higenbottam TW. A simultaneous single breath measurement of pulmonary diffusing capacity with nitric oxide and carbon monoxide. Eur Respir J. 1989 Jan;2(1):56-63. PMID 2707403
- [Background] Wemeau-Stervinou L, Perez T, Murphy C, Polge AS, Wallaert B. Lung capillary blood volume and membrane diffusion in idiopathic interstitial pneumonia. Respir Med. 2012 Apr;106(4):564-70. doi: 10.1016/j.rmed.2011.12.011. Epub 2012 Jan 4. PMID 22221584
- [Derived] Barisione G, Brusasco C, Garlaschi A, Baroffio M, Brusasco V. Lung diffusing capacity for nitric oxide as a marker of fibrotic changes in idiopathic interstitial pneumonias. J Appl Physiol (1985). 2016 May 1;120(9):1029-38. doi: 10.1152/japplphysiol.00964.2015. Epub 2016 Feb 18. PMID 26893034